CLINICAL TRIAL: NCT00065754
Title: Brain Imaging and Pain: Analysis of Placebo Analgesia
Brief Title: Brain Imaging and Pain in Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double
Other Study IDs: R01AT001424-01 (NIH); R01AT001424-01 (NIH)
Record Dates: First submitted 2003-07-31; First posted 2003-08-01 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-08

CONDITIONS: Irritable Bowel Syndrome
Keywords: Placebo; Analgesia; Pain; Brain mechanism; Expectation
MeSH Terms: conditions — Irritable Bowel Syndrome; Agnosia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: placebo

SUMMARY:
This study examines the mechanisms, including brain imaging of placebo analgesia

ELIGIBILITY:
Inclusion criteria:

* Irritable Bowel Syndrome
* English speaking

Exclusion criteria:

* Chronic pain condition other than Irritable Bowel Syndrome
* Medical condition that would contraindicate use of lidocaine
* Clinical criteria for fibromyalgia
* Presence of systemic disease such as diabetes, thyroid, gastrointestinal or liver disease, collagen vascular disease, malignancy, focal or neurological
* Seropositive HIV
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Robinson, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States